CLINICAL TRIAL: NCT05612659
Title: Developing an EEG Probe for Studying Effects of Non-invasive Cortical and Spinal Cord Electrical Stimulation on Cognitive Control in Post Stroke Depression
Brief Title: Developing an EEG Probe for Studying and Modulating Cognitive Control
Acronym: PSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Ishita Basu, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EEG_noninvasive_stimulation
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Post-stroke Depression
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Electrical stimulation (Experimental): Subjects will receive transcranial electrical stimulation.
  Interventions: Procedure: Transcranial Electrical stimulation
- Transcutaneous direct current stimulation (Experimental): Subjects will receive Transcutaneous direct current stimulation
  Interventions: Procedure: Transcutaneous direct current stimulation

INTERVENTIONS:
Procedure: Transcranial Electrical stimulation — Noninvasive electrical stimulation of lateral frontal cortex.
  Arms: Transcranial Electrical stimulation
Procedure: Transcutaneous direct current stimulation — Noninvasive electrical stimulation of the T10 spinal column.
  Arms: Transcutaneous direct current stimulation

SUMMARY:
This study aims to investigate effects of transcranial current stimulation (tES) and transcutaneous direct current stimulation (tsDCS) associated changes on fronto-parietal EEG and cognitive performance in patients with post stroke depression (PSD)

DETAILED DESCRIPTION:
The investigators will perform a double blind, randomized, sham controlled, crossover study design to assess effects of tES, tsDCS and sham stimulation on the performance during a cognitive control task. The working Hypothesis is tsDCS and/or tES will enhance frontal theta oscillations as recorded on EEGs and improve task performance compared to sham stimulation.

Results from this project can potentially lead to the development of a new research tool for assessing neuromodulation strategies to treat mental disorders and their comorbidities. It will also uncover the neural correlates of cognitive deficits in PSD and provide feasible biomarkers associated with treatment response in support of a larger clinical.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will include both male and female of age over 18 years and a BMI of 18-35 Kg/mts2 who have experienced stroke.
2. Moderately depressed, MADRS:18-28, PHQ9: 10-20 and/or experiencing cognitive impairments after stroke

Exclusion Criteria:

1. Current or lifetime bipolar disorder or schizophrenia diagnosis;
2. current (past month): PTSD, psychotic or substance use disorder (nicotine and caffeine allowed);
3. significant risk of suicide according to CSSRS or clinical judgment, or suicidal behavior in the past year:
4. current chronic severe pain conditions;
5. current chronic use of: opioids analgesics, medications that affect blood pressure or drugs with significant autonomic effects (stimulants and antipsychotics allowed if dose stable for 1 month);
6. skin lesions on electrode placement region;
7. implanted electrical medical devices;
8. Pregnancy;
9. suspected IQ<80, and 10) any other clinically relevant reason as judged by the clinician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
EEG oscillations | change from baseline
  Theta (4-8 Hz) oscillations in the mid frontal EEG

SECONDARY OUTCOMES:
Behavior | during procedure
  Response time in a multi source interference task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided